CLINICAL TRIAL: NCT02107729
Title: The Importance of Needle Gauge for Pain During Injection of Local Anaesthetic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/2297B
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Needlestick Injuries
Keywords: Injections; Pain; Healthy volunteers; Lidocaine
MeSH Terms: conditions — Needlestick Injuries; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Needle gauge small (Experimental): injection needle 23 G
  Interventions: Procedure: Large needle gauge lidocaine injection; Procedure: Normal needle gauge lidocaine injection; Procedure: Small needle gauge lidocaine injection
- Needle gauge normal (Experimental): injection needle 25 G
  Interventions: Procedure: Large needle gauge lidocaine injection; Procedure: Normal needle gauge lidocaine injection; Procedure: Small needle gauge lidocaine injection
- Needle gauge large (Experimental): injection needle 27 G
  Interventions: Procedure: Large needle gauge lidocaine injection; Procedure: Normal needle gauge lidocaine injection; Procedure: Small needle gauge lidocaine injection

INTERVENTIONS:
Procedure: Large needle gauge lidocaine injection — 21 G
Procedure: Normal needle gauge lidocaine injection — 23 G
Procedure: Small needle gauge lidocaine injection — 27 G

SUMMARY:
This study will investigate the influence of needle gauge on pain during injection of local anaesthetic. Healthy volunteers will be recruited, who will each receive three injections with either 21G, 23G or 27G subcutaneously on the abdomen. After each injection, the participants will be asked to evaluate the pain on a Visual analog scale (0-100 mm). It is anticipated that the pain will decrease with decreasing thickness of the needle. The aim of this study is to find a simple method for pain reduction that can be used in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years

Exclusion Criteria:

* Kidney, heart or liver disease
* Eczema or psoriasis on injection site
* Neuropathy
* Regular use of painkillers
* Hypersensitivity of Lidocaine
* Pregnancy
* Diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Pain | 60 seconds
  1. Visual analog scale
  2. Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vilhjalmur Finsen, Prof md, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of Neuroscience, NTNU, Trondheim, Norway

REFERENCES:
- [Result] Wago KJ, Skarsvag TI, Lundbom JS, Tangen LF, Ballo S, Hjelseng T, Finsen V. The importance of needle gauge for pain during injection of lidocaine. J Plast Surg Hand Surg. 2016;50(2):115-8. doi: 10.3109/2000656X.2015.1111223. Epub 2015 Nov 23. PMID 26595751